CLINICAL TRIAL: NCT06887231
Title: Virtual Reality (VR) Platform and Transcutaneous Electrical Nerve Stimulation (TENS) for Early Stroke Rehabilitation
Brief Title: Virtual Reality and Neurostimulation for Early Stroke Rehabilitation
Acronym: VR-TENS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Stanisa Raspopovic, Professor, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2280/2024
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Stroke
Keywords: Stroke; Virtual Reality; Transcutaneous Electrical Nerve Stimulation; Multisensory integration; Task oriented movement; Rehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR+TENS (Experimental): Patients will engage in goal-directed upper-limb rehabilitation exercises within a virtual reality environment. During these exercises, they will receive synchronized electrical stimulation targeting the median nerve.
  The intervention phase will span three weeks, with patients participating in at least three sessions per week, each lasting approximately 60 minutes.
  Interventions: Other: VR+TENS
- Conventional Rehabilitation (Active Comparator): Participants will undergo the same therapy duration, engaging in conventional physiotherapy, occupational therapy, or physical therapy. Exercises and movements will be designed to align with those in the experimental group.
  Interventions: Other: Conventional rehabilitation

INTERVENTIONS:
Other: VR+TENS — Patients will perform task-oriented movements in an immersive scenario while receiving congruent electrical stimulation. During each session, multiple games will be played, with the type and difficulty calibrated based on the patient's level of impairment.
  Arms: VR+TENS
Other: Conventional rehabilitation — Patients will perform dose-matched conventional rehabilitation (aligned with the intervention group), which will include physiotherapy, occupational therapy, and physical therapy.
  Arms: Conventional Rehabilitation

SUMMARY:
Stroke is one of the leading causes of disability, leaving millions of individuals each year impaired with lasting motor and sensory impairments. In the subacute phase, which goes from the first week to 3 months post-stroke, the patient has the highest recovery, which could be boosted by proper technologies intended for the rehabilitation of the patients. The impairments that the patients experience are extremely heterogeneous and go from muscle weakness to spasticity of the paretic side of the body. Beyond motor deficits, stroke survivors also suffer from sensory impairment (they do not properly feel with the paretic side of their body), impaired body representation (misjudging the size, position, and movement of their affected limb), which can further hinder recovery.

Traditional rehabilitation primarily targets motor function, often without considering at all the role of sensory feedback and body perception in the recovery process. However, growing evidence suggests that the combination of multiple sensory modalities towards a multifaceted rehabilitation can enhance neuroplasticity and improve rehabilitation outcomes.

To address this, the investigators have developed a novel rehabilitation approach that integrates immersive virtual reality (VR) with transcutaneous electrical nerve stimulation (TENS). This system allows stroke patients to interact with a virtual environment while receiving synchronized tactile stimulation, reinforcing sensorimotor integration. Unlike conventional therapy, which relies on passive or repetitive exercises, this approach engages patients in active, goal-oriented movements, tailored to their individual recovery progress.

By focusing on the subacute stroke population, this project aims to leverage the brain's heightened plasticity during early recovery to maximize functional improvements. The VR-based intervention will adapt to each patient's motor abilities, providing real-time feedback to encourage precise movements and enhance sensory processing. Through this multisensory experience, the investigators seek to improve not only motor control but also sensory and body representation measures.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of ischemic or hemorrhagic stroke
* In the subacute phase (from 7 days to 3 months from last stroke onset)
* Fugl-Meyer-Upper Extremity (FMUE) scale for the motor part: FMUE ≥ 10
* Ability to sit in an upright position
* Age between 18 and 80 years

Exclusion Criteria:

* Other neurological or physical impairment or mental condition that, in the judgment of the investigator, does not allow participation in the study.
* Mini-Mental State Examination (MMSE) < 24
* Epilepsy
* Nausea, headaches or fatigue due to VR-generated environment ("virtual reality motion sickness")
* Peripheral nerve damage in the affected arm or hand
* Pacemaker or other electronic implants

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Changes in functional performances | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To assess functional performance of the upper extremity through observational means the investigators will use the Action Research Arm Test (ARAT). The ARAT is a 19-item measure divided into 4 sub-tests (grasp, grip, pinch, and gross arm movement). The total score goes from 0 to 57. Performance on each item is rated on a 4-point ordinal scale ranging from: 3) Performs test normally 2) Completes test, but takes abnormally long or has great difficulty 1) Performs test partially 0) Can perform no part of test.
Changes in sensorimotor impairments | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To assess the sensorimotor impairment in individuals who have had a stroke the investigators will use Fugl-Meyer for upper extremity (FMUE). FMUE assesses reflex activity, movement control, muscle strength, and sensory performances. It comprises items scored on a scale of 0 to 2, where 0 = cannot perform, 1 = performs partially and 2 = performs fully.
Changes in upper limb body representation | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure the body representation of the subjects the investigators will use body-landmark metric. In VR, the subject is asked to locate the position of specific body landmarks (e.g. elbow, inner wrist, outer wrist, index, ring) describing the proportion of patients' arm while a black panel is on top of his/her arm. The investigators will then compare the real and perceived dimension of patients' arm

SECONDARY OUTCOMES:
Changes in degree of assistance required | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To assess the degree of assistance required by an individual on ten mobility and self-care the investigators will use the Barthel Index. The score goes from 0 to 100. It consists of an ordinal scale which measures a person's ability to complete activities of daily living (ADL)
Changes in spasticity at hand and elbow level | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  The investigators will use Modified Ashworth Scale to test resistance to passive movement about a joint with varying degrees of velocity. This test is performed by extending the patients limb first from a position of maximal possible flexion to maximal possible extension (the point at which the first soft resistance is met).
Changes in peripersonal space | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure the peri-personal space of stroke patients (the space in which multisensory integration is enhanced). Test Performance: In VR, the subject is sitting on a table and sees balls approaching him. He/she's asked to press a controller whenever he/she feels electrical stimulation.
Changes in tactile acuity | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure the tactile acuity of patients we will use the Two-Point discrimination test. While blindfolded, the patient is repetitively touched with either one or two pins (fixed distance) and he asked to tell how many pins he/she feels.
Changes in spatial neglect (CBS) | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure spatial neglect, participants will be assessed using the Catherine Bergego Scale, which comprises 10 everyday tasks observed during self-care activities. A therapist scores the patient on behaviors such as neglecting the left side of the body and difficulties in grooming, eating, movement, and spatial awareness. The CBS uses a 4-point scale (0-3) to rate neglect severity, with a total score of 30.
Changes in spatial neglect (LBT) | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To measure spatial neglect, patients will perform a line bisection test. The Line Bisection Test is a test is a quick measure to detect the presence of unilateral spatial neglect (USN). To complete the test, one must place a mark with a pencil through the center of a series of horizontal lines. Usually, a displacement of the bisection mark towards the side of the brain lesion is interpreted as a symptom of neglect.
Changes in upper limb kinematics (Velocity) | Every day, from day 1 to day 14
  To assess changes in velocity the investigators will measure kinematic velocity of the patients while performing rehabilitation tasks.
Changes in upper limb kinematics (Smoothness) | Every day, from day 1 to day 14
  To assess changes in smoothness the investigators will measure kinematic smoothness of the patients while performing rehabilitation tasks.
Changes in upper limb kinematics (Efficiency) | Every day, from day 1 to day 14
  To assess changes in efficiency the investigators will measure the amount and rate of task-oriented movements of the patients.
Changes in upper limb kinematics (Precision) | Every day, from day 1 to day 14
  To assess changes in precision the investigators will measure the spatial precision (error with respect to a predefined correct movement) during the task-oriented movements of the patient.

OTHER OUTCOMES:
Changes in pain | day 0 (before the first rehabilitation session, T0); 1.5 week (after six rehabilitation sessions, T1); 3 weeks (one day after the last rehabilitation session, T2); 5 weeks (2 weeks after the last rehabilitation session,T3)
  To quantify the experience of pain. This will be evaluated with Visual Analogue Scale (VAS). The score goes from 0 to 10 where 0 means no pain and 10 means the worst possible pain.
Treatment Satisfaction | 3 weeks (one day after the last rehabilitation session, T2)
  To assess treatment satisfaction, participants will complete the Treatment Satisfaction Questionnaires, rated on a scale from 0 to 10 where 0 means complete dissatisfaction and 10 means maximum satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Department of Neurology, Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fugl-Meyer AR, Jaasko L, Leyman I, Olsson S, Steglind S. The post-stroke hemiplegic patient. 1. a method for evaluation of physical performance. Scand J Rehabil Med. 1975;7(1):13-31. PMID 1135616
- [Background] Aurucci GV, Gozzi N, Wagner M, Preatoni G, Brunello N, Cimolato A, Secerovic N, Zipser CM, Raspopovic S. Targeted neural stimulation congruent with immersive reality decreases neuropathic pain. Brain Stimul. 2025 Sep-Oct;18(5):1671-1674. doi: 10.1016/j.brs.2025.08.023. Epub 2025 Aug 29. No abstract available. PMID 40886914
- [Background] Aurucci GV, Preatoni G, Damiani A, Raspopovic S. Brain-Computer Interface to Deliver Individualized Multisensory Intervention for Neuropathic Pain. Neurotherapeutics. 2023 Sep;20(5):1316-1329. doi: 10.1007/s13311-023-01396-y. Epub 2023 Jul 5. PMID 37407726
- [Background] Bolognini N, Russo C, Edwards DJ. The sensory side of post-stroke motor rehabilitation. Restor Neurol Neurosci. 2016 Apr 11;34(4):571-86. doi: 10.3233/RNN-150606. PMID 27080070
- [Background] Perez-Marcos D. Virtual reality experiences, embodiment, videogames and their dimensions in neurorehabilitation. J Neuroeng Rehabil. 2018 Nov 26;15(1):113. doi: 10.1186/s12984-018-0461-0. PMID 30477527
- [Background] Hao J, He Z, Yu X, Remis A. Comparison of immersive and non-immersive virtual reality for upper extremity functional recovery in patients with stroke: a systematic review and network meta-analysis. Neurol Sci. 2023 Aug;44(8):2679-2697. doi: 10.1007/s10072-023-06742-8. Epub 2023 Mar 23. PMID 36959332
- [Background] Laver KE, Lange B, George S, Deutsch JE, Saposnik G, Crotty M. Virtual reality for stroke rehabilitation. Cochrane Database Syst Rev. 2017 Nov 20;11(11):CD008349. doi: 10.1002/14651858.CD008349.pub4. PMID 29156493
- [Background] Chen Y, Abel KT, Janecek JT, Chen Y, Zheng K, Cramer SC. Home-based technologies for stroke rehabilitation: A systematic review. Int J Med Inform. 2019 Mar;123:11-22. doi: 10.1016/j.ijmedinf.2018.12.001. Epub 2018 Dec 11. PMID 30654899
- [Background] A. Serino et al., 'Peripersonal Space: An Index of Multisensory Body-Environment Interactions in Real, Virtual, and Mixed Realities', Front. ICT, vol. 4, Jan. 2018, doi: 10.3389/fict.2017.00031.
- [Background] Crema A, Bassolino M, Guanziroli E, Colombo M, Blanke O, Serino A, Micera S, Molteni F. Neuromuscular electrical stimulation restores upper limb sensory-motor functions and body representations in chronic stroke survivors. Med. 2022 Jan 14;3(1):58-74.e10. doi: 10.1016/j.medj.2021.12.001. Epub 2022 Jan 7. PMID 35590144
- [Background] Bassolino M, Franza M, Guanziroli E, Sorrentino G, Canzoneri E, Colombo M, Crema A, Bertoni T, Mastria G, Vissani M, Sokolov AA, Micera S, Molteni F, Blanke O, Serino A. Body and peripersonal space representations in chronic stroke patients with upper limb motor deficits. Brain Commun. 2022 Aug 5;4(4):fcac179. doi: 10.1093/braincomms/fcac179. eCollection 2022. PMID 35950092
- [Background] Mastria G, Bertoni T, Perrin H, Akulenko N, Risso G, Akselrod M, Guanziroli E, Molteni F, Hagmann P, Bassolino M, Serino A. Body ownership alterations in stroke emerge from reduced proprioceptive precision and damage to the frontoparietal network. Med. 2025 Apr 11;6(4):100536. doi: 10.1016/j.medj.2024.10.013. Epub 2024 Nov 11. PMID 39532102
- [Background] Matamala-Gomez M, Malighetti C, Cipresso P, Pedroli E, Realdon O, Mantovani F, Riva G. Changing Body Representation Through Full Body Ownership Illusions Might Foster Motor Rehabilitation Outcome in Patients With Stroke. Front Psychol. 2020 Aug 21;11:1962. doi: 10.3389/fpsyg.2020.01962. eCollection 2020. PMID 32973612
- [Background] Takeuchi N, Izumi S. Maladaptive plasticity for motor recovery after stroke: mechanisms and approaches. Neural Plast. 2012;2012:359728. doi: 10.1155/2012/359728. Epub 2012 Jun 26. PMID 22792492
- [Background] Doyle S, Bennett S, Fasoli SE, McKenna KT. Interventions for sensory impairment in the upper limb after stroke. Cochrane Database Syst Rev. 2010 Jun 16;2010(6):CD006331. doi: 10.1002/14651858.CD006331.pub2. PMID 20556766
- [Background] Langhorne P, Bernhardt J, Kwakkel G. Stroke rehabilitation. Lancet. 2011 May 14;377(9778):1693-702. doi: 10.1016/S0140-6736(11)60325-5. PMID 21571152
- [Background] Lucas-Noll J, Clua-Espuny JL, Lleixa-Fortuno M, Gavalda-Espelta E, Queralt-Tomas L, Panisello-Tafalla A, Carles-Lavila M. The costs associated with stroke care continuum: a systematic review. Health Econ Rev. 2023 May 17;13(1):32. doi: 10.1186/s13561-023-00439-6. PMID 37193926
- [Background] Strilciuc S, Grad DA, Radu C, Chira D, Stan A, Ungureanu M, Gheorghe A, Muresanu FD. The economic burden of stroke: a systematic review of cost of illness studies. J Med Life. 2021 Sep-Oct;14(5):606-619. doi: 10.25122/jml-2021-0361. PMID 35027963
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] He Q, Wang W, Zhang Y, Xiong Y, Tao C, Ma L, Ma J, You C, Wang C. Global, Regional, and National Burden of Stroke, 1990-2021: A Systematic Analysis for Global Burden of Disease 2021. Stroke. 2024 Dec;55(12):2815-2824. doi: 10.1161/STROKEAHA.124.048033. Epub 2024 Oct 17. PMID 39417225
- [Background] Lang CE, Wagner JM, Dromerick AW, Edwards DF. Measurement of upper-extremity function early after stroke: properties of the action research arm test. Arch Phys Med Rehabil. 2006 Dec;87(12):1605-10. doi: 10.1016/j.apmr.2006.09.003. PMID 17141640